CLINICAL TRIAL: NCT00528216
Title: A Randomized, Controlled, Single-Blind Study to Investigate the Effect of Three Capsaicin Dermal Liquid Formulations on Epidermal Nerve Fiber Immunostaining and Sensory Function In Healthy Volunteers
Brief Title: Study of Three Capsaicin Dermal Liquid Formulations on Epidermal Nerve Fiber Immunostaining and Sensory Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeurogesX (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: C201
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-03

CONDITIONS: Pain
Keywords: Analgesics; Capsaicin
MeSH Terms: conditions — Pain

INTERVENTIONS:
Drug: Capsaicin Dermal Liquid

SUMMARY:
The purpose of this study is to evaluate potential changes in epidermal nerve fiber immunostaining (ENFI) and sensory nerve function in healthy normal volunteers following single applications of three different investigational topical Capsaicin Dermal Liquids (10% w/v trans capsaicin), and a comparable control (propylene glycol). In addition, the pain and tolerability of the application of each formulation will also be assessed. Data from this clinical study may be used to select a formulation for further clinical evaluation.

DETAILED DESCRIPTION:
This is a randomized, controlled, single-blind, single-center, Phase 1 study in twenty normal healthy volunteers. Each subject will have a single 15 minute exposure to each of three topical Capsaicin Dermal Liquids and the control. Each application site, located on the distal and proximal anterior medial thigh areas, will be 5.0 × 5.0 cm in size. The volume applied will be 15 mcL per cm2 and hence the total volume applied will be 375 mcL.

At baseline and prior to skin punch biopsy at Day 7, QST of the four application sites for warming and cooling detection thresholds, and assessment of mechanical (sharp pain) sensation and tactile thresholds, will be performed and evaluated. This will be repeated at each of the four application sites on Day 7 and the Termination Visit.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years of age.
* Be in good health.
* Have intact, unscarred skin over the thighs.
* Agree not to use topically-applied products containing non-steroidal anti-inflammatory drugs, menthol, methyl salicylate, other counterirritants, local anesthetics, steroids or capsaicin anywhere on the thighs for the duration of the study.
* Female subjects must not be breast-feeding and must have a negative serum beta human chorionic gonadotropin (hCG) pregnancy test performed within 7 days prior to the Application Visit (Day 0).
* All subjects, including early terminations, must be willing to use effective methods of birth control and/or refrain from participating in a conception process during the study and for 30 days following experimental drug exposure.
* Subjects must be willing and able to comply with protocol requirements for the duration of study participation. Requirements include but are not limited to attending all study visits and refraining from extensive travel during study participation.
* Subjects must sign an informed consent form for this study approved by the Investigator's Institutional Review Board (IRB).

Exclusion Criteria:

* Any dermatological condition(s) that in the judgment of the Principal Investigator has the potential to disrupt skin integrity or alter sensory function on the thighs.
* Any skin infection, skin irritation (e.g., poison oak), history of eczema, trauma or burn (including sunburn) on the thighs within 30 days preceding the Application Visit (Day 0).
* Any medical history of painful conditions, surgery, or injury involving or affecting the thighs, including but not limited to prior orthopedic surgery, lumbrosacral disc disease, sciatica, and hip or femur fracture.
* Any medical history of known or suspected body system abnormalities, including but not limited to diabetes, hypothyroidism, asthma or any form of peripheral or central nervous system disease.
* Use of any systemic medications that interact with the peripheral nervous system, including beta adrenergic blockers, alpha adrenergic blockers, anticonvulsant drugs, antidepressant drugs or opioids within 30 days prior to the Application Visit (Day 0).
* Use of any topically-applied product including prescription or over the-counter (OTC) analgesic creams/lotions/patches, non steroidal anti-inflammatory drugs, counterirritants, local anesthetics, steroids or capsaicin on the thighs within 30 days preceding the Application Visit (Day 0).
* Currently taking any prescription medication except for oral, transdermal or injected contraceptives.
* Requirement for ongoing or periodic pain medication for any chronic or recurrent medical condition.
* Participation in another drug research study within 30 days preceding the Application Visit (Day 0).
* Diagnosis of human immunodeficiency virus (HIV) infection, according to medical history and/or self-report.
* History or current substance abuse including alcoholism/alcohol abuse, as judged by the investigator.
* Positive test result on the urine drug screen for opioids, cannabis, phencyclidine (PCP), cocaine and amphetamines performed at the Screening Visit.
* History of hypersensitivity to capsaicin (i.e., chili peppers or OTC capsaicin products), local anesthetics (including lidocaine), adhesives or any other components (see Table 2) of the formulations.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Tobias, MD, Study Director — NeurogesX